CLINICAL TRIAL: NCT00652405
Title: Effect of Moderate Alcohol Consumption on Cephalic Phase Reflex and Gene Expression of Adipose Tissue in Postmenopausal Women
Brief Title: Effect of Alcohol on Cephalic Phase Reflex and Gene Expression
Acronym: AR22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Responsible Party: Henk Hendriks, TNO Quality of Life
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: P8009
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2008-05

CONDITIONS: Type 2 Diabetes; Inflammation; Carbohydrate&Lipid Metabolism; Oral Processing
Keywords: cephalic phase reflex; gene expression; inflammation; adiponectin; pancreatic polypeptide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment A (Experimental): four weeks of white wine consumption (25g alcohol/day; ~2.5 standard drinks)
  Interventions: Dietary Supplement: alcohol
- Treatment B (Placebo Comparator): Four weeks of water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: alcohol — 250 ml of white wine (13% vol; ~25 gram of alcohol per day)
  Arms: treatment A
Dietary Supplement: Placebo — 250 ml of mineral water (Brand name: Vittel)
  Arms: Treatment B

SUMMARY:
Moderate alcohol consumption has consistently been associated with lowered risk of developing type two diabetes mellitus compared to abstainers and heavy drinkers. However, the underlying mechanism for the lower risk of type two diabetes is not clear.

Hypothesis: moderate alcohol consumption for four weeks changes gene expression pathways of inflammatory status, insulin sensitivity and lipid and carbohydrate metabolism in adipose tissue in both lean and obese postmenopausal women.

Hypothesis: Oral sensory stimulation by means of alcohol in the oral cavity will induce a cephalic phase reflex as indicated by increased autonomic & endocrine responses in postmenopausal women.

DETAILED DESCRIPTION:
Moderate alcohol consumption has consistently been associated with lowered risk of developing type two diabetes mellitus compared to abstainers and heavy drinkers. However, the physiological mechanism for this is not known.

Two potential mechanisms will be investigated in this study to explain the findings from observational studies: One concerning more acute changes upon alcohol consumption (cephalic phase reflex) which could explain the observed improvement in postprandial glycemia after alcohol consumption; the other has to do with metabolic changes after more prolonged moderate alcohol consumption in gene expression of adipose tissue which might lead to improved insulin sensitivity. Both mechanisms will be discussed below.

Cephalic phase reflex Mere exposure to smell, sight, taste and textural attributes of foods elicits myriad digestive, endocrinologic, thermogenic, cardiovascular and renal responses. These responses are rapid (generally occurring in minutes of sensory stimulation), small (relative to the magnitude achieved when food is actually being metabolized) and transient (retuning to baseline levels within minutes). They are termed pre-absorptive or cephalic phase reflexes/responses (CPR) and refer to a set of food intake-associated autonomic and endocrine responses to the stimulation of sensory systems mainly located in the oropharyngeal cavity. Their function may be essential adaptive, preparing the digestive system for the reception, digestion and absorption of ingested nutrients.

The release of cephalic phase hormones occurs through activation of vagal efferent fibers in response to food-related sensory stimuli. Pancreatic polypeptide (PP) is a hormone almost exclusively under vagal control increases. Thus, the cephalic phase PP response is a sensitive indicator of vagal activation to food stimuli. PP levels rise up to 100% above baseline when individuals taste, chew and expectorate food while the magnitude of cephalic phase insulin release is relatively small (25% above baseline). The cephalic phase is by some considered as a reflex rather then a response as it is dependent on neural rather than nutrient-induced stimulation.

The physiological significance of the cephalic phase hormonal responses is demonstrated by experimental manipulations which inhibit or bypass cephalic phase insulin release. Under these circumstances, hyperglycemia and hyperinsulinemia are evident.

Alcohol consumption lowers postprandial glucose concentrations and improves insulin secretion. Furthermore, alcohol consumption increases postprandial diet-induced thermogenesis, heart rate and causes diuresis presumably resulting from inhibition of vasopressin. Since in the postprandial state, almost all cephalic phase responses are affected by alcohol, it seems plausible that the human body might exhibit a CPR upon oral sensory stimulation by alcohol-containing beverages. This study therefore investigates for the first time if and to what extent alcohol triggers CPR which may account for the improved postprandial glycemia seen after alcohol consumption.

Gene expression in adipose tissue Application of transcriptomics technology, via gene expression profiling, with the use of microarrays is a powerful but expensive tool for identifying molecular pathways responsible for metabolic regulation. Gene expression profiling in human intervention studies, allows for genome wide screening of the effects of specific diets or nutrients and results in biomarker profiles. Recently, it has been used to detect new important signaling pathways involved in glucose and lipid metabolism.

Adipose tissue has important metabolic and endocrine functions. Changes in these functions are associated with an increased low-grade inflammatory state and with chronic diseases such as obesity and diabetes. Furthermore, changes in gene expression profiles of subcutaneous adipose tissue can be observed after nutritional interventions.

An important hormone almost exclusively and abundantly secreted by adipose tissue is adiponectin. Circulating adiponectin levels in lean persons are far above any other hormone. It is believed that these high levels of adiponectin protect lean persons while its decrease in obesity is associated with a low grade inflammation and the development of insulin resistance and diabetes. Research by our group has shown that moderate alcohol consumption increases both plasma levels and mRNA adiponectin levels. This suggests that moderate alcohol consumption, directly or indirectly, exerts effects on adipose tissue gene expression. Since adiponectin is associated with inflammatory status, lipid metabolism and insulin sensitivity, changes in gene expression of these pathways are expected after alcohol consumption to be reflected in adipose gene expression.

Beneficial effects of moderate alcohol consumption might be more apparent in lean then in overweight persons. Compared to overweight men, lean men have stronger increases in adiponectin and in the 'good' HDL cholesterol after moderate alcohol consumption. Furthermore, liver enzymes of obese subjects are elevated after moderate alcohol consumption indicating a less favorable response to moderate alcohol consumption among overweight persons. Since the current rise in the obesity pandemic, different responses between lean and obese subjects after alcohol consumption are of great importance.

Thus, investigating alcohol-induced changes in gene expression of adipose tissue in both lean and overweight subjects could not only be highly valuable for the identification of new biomarkers but could also be of pivotal importance to identify specific physiological mechanisms leading to improved insulin sensitivity and reduced inflammatory status. This eventually could help in the general understanding of the development of diet-related chronic disorders such as obesity and type two diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the health and lifestyle questionnaire (P8009 F02), physical examination and results of the pre-study laboratory tests
2. Caucasian postmenopausal females aged 65 years or younger at Day 01 of the study.
3. Body Mass Index (BMI) of 18 - 26 or 27 - 35 kg/m2.
4. Postmenopausal as assessed by self reported absence of menstrual periods for at least 12 months.
5. Alcohol consumption ≥ 5 and ≤ 22 standard units/week.
6. Normal Dutch eating habits as assessed by P8009 F02.
7. Voluntary participation.
8. Having given written informed consent.
9. Willing to comply with the study procedures, including refrain from drinking alcoholic drinks other then the wine provided by TNO during the entire study.
10. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years.
11. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study.
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances.
3. Having a history of medical or surgical events that may significantly affect the study outcome, particularly metabolic or endocrine disease and gastrointestinal disorders.
4. Use of medication that may affect the outcome of the study parameters.
5. Having a family history of alcoholism.
6. Smoking.
7. Not having appropriate veins for blood sampling/cannula insertion according to TNO.
8. Reported unexplained weight loss or gain in the month prior to the pre-study screening.
9. Reported slimming or medically prescribed diet.
10. Reported vegan, vegetarian or macrobiotic.
11. Recent blood donation (<1 month prior to the start of the study).
12. Not willing to give up blood donation during the study.
13. Personnel of TNO Quality of Life, their partner and their first and second degree relatives.
14. Not having a general practitioner.
15. Not willing to accept information transfer concerning participation in the study, or information regarding her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.
16. Not willing your general practitioner to be notified upon participation in this study

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Gene expression profiles in adipose tissue | after four weeks of intervention
Pancreatic Polypeptide (PP) | 0, 4, 8, 12, 16, 20 and 30 min after start of modified sham-feeding with either water, white wine or cake

SECONDARY OUTCOMES:
Cytokines excreted from PBMCs after in vitro stimulation with LPS | after four weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Henk FJ Hendriks, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Netherlands

REFERENCES:
- [Result] Joosten MM, Balvers MG, Verhoeckx KC, Hendriks HF, Witkamp RF. Plasma anandamide and other N-acylethanolamines are correlated with their corresponding free fatty acid levels under both fasting and non-fasting conditions in women. Nutr Metab (Lond). 2010 Jun 14;7:49. doi: 10.1186/1743-7075-7-49. PMID 20546561
- [Result] Joosten MM, de Graaf C, Rietman A, Witkamp RF, Hendriks HF. Short-term oral exposure to white wine transiently lowers serum free fatty acids. Appetite. 2010 Aug;55(1):124-9. doi: 10.1016/j.appet.2010.04.217. Epub 2010 May 11. PMID 20438782